CLINICAL TRIAL: NCT06186037
Title: Clinical Comparison of Low-dose Rosuvastatin Plus Ezetimibe Combination Therapy and High-dose Rosuvastatin Monotherapy in Patients With Minimal to Intermediate Coronary Artery Disease Without Percutaneous Coronary Intervention : A Prospective, Multicenter, Randomized, Open-label Trial
Brief Title: Clinical Comparison of Low-dose Rosuvastatin Plus Ezetimibe Combination Therapy and High-dose Rosuvastatin Monotherapy in Patients With Minimal to Intermediate Coronary Artery Disease Without Percutaneous Coronary Intervention
Acronym: ALMIGHTY
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Saint Vincent's Hospital, Korea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XC23MIDV0033
Record Dates: First submitted 2023-11-21; First posted 2023-12-29 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Disease; Dyslipidemias; Primary Prevention
Keywords: Coronary Artery Disease; Dyslipidemias; Primary Prevention
MeSH Terms: conditions — Coronary Artery Disease; Dyslipidemias | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination drug group of Ezetimibe 10 mg/Rosuvastatin 5 mg (Experimental): Ezetimibe 10 mg/Rosuvastatin 5 mg, Oral administration once a day, taking it for 3 years
  Interventions: Drug: Combination drug group of Ezetimibe 10 mg/Rosuvastatin 5 mg
- Mono drug group of Rosuvastatin 20 mg (Active Comparator): Rosuvastatin 20 mg , Oral administration once a day, taking it for 3 years
  Interventions: Drug: Mono drug group of Rosuvastatin 20 mg

INTERVENTIONS:
Drug: Combination drug group of Ezetimibe 10 mg/Rosuvastatin 5 mg — Oral administration once a day, taking it for 3 years
  Arms: Combination drug group of Ezetimibe 10 mg/Rosuvastatin 5 mg
Drug: Mono drug group of Rosuvastatin 20 mg — Oral administration once a day, taking it for 3 years
  Arms: Mono drug group of Rosuvastatin 20 mg

SUMMARY:
[Purpose of the Clinical Study]:The purpose of this study is to conduct a clinical comparison of low-dose rosuvastatin plus ezetimibe combination therapy and high-dose rosuvastatin monotherapy in patients with minimal to intermediate coronary artery disease without percutaneous coronary intervention to confirm non-inferiority in the reduction of key cardiovascular events.

[Hypothesis]:In patients who have not undergone percutaneous coronary intervention for minimal to moderate coronary artery disease, low-dose rosuvastatin and ezetimibe combination therapy are non-inferior in terms of reducing major cardiovascular events compared to high-dose rosuvastatin monotherapy.

DETAILED DESCRIPTION:
[Background]:While high-dose statin is becoming more important, there are factors that limit more widespread use of such a treatment due to the possibility of adverse events, especially among the patients from East Asia. These factors include muscle-related diseases, higher liver figures, and onset of diabetes. Meanwhile, the combination treatment of low-dose statin and ezetimibe, which slows down the absorption of LDL cholesterol, can see an equivalent level of LDL cholesterol reduction compared to high-dose statin treatments, while having an advantage in terms of the level of decrease in adverse events. However, further verification is still needed whether the statin + ezetimibe combination therapy and the high-dose statin monotherapy of the same reduction effect against LDL cholesterol would have the same level of clinical utility. Especially with regard to the treatment of patients with minimal to minor coronary artery diseases, there are no available guidelines for the use of statin. In the case of a stenosis lesion with a 50 to 70% severity level, the likelihood of choosing medication over percutaneous coronary artery interventions through a physiological evaluation is increasing compared to the past. Also, some studies suggested that the MACE of an intermediate lesion showed a difference depending on the administration of statin, while percutaneous coronary intervention did not. Therefore, verification of the clinical utility on the said lesions is also necessary.

[Clinical Research Plan]: A prospective, multicenter, randomized, and public label clinical study involving a total of 6,356 patients, 3,178 patients each with ezetimibe 10mg/rosuvastatin 5mg (experimental group) and rosuvastatin 20mg (active control group), in patients who have not undergone percutaneous coronary intervention for minimal to moderate coronary artery disease. After random assignment, take the assigned drugs for 3 years and follow-up observation is conducted at 6weeks, 6, 12, and 36 months. Test personnel can follow up through hospital visits or phone visits. The primary end-points are a combined assessment variable of all cause death, cardiovascular deaths, myocardial infarction without death, stroke without death, hospitalization due to unstable angina, and revascularization after random assignment at 36 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adjusts (19 or older)
2. Patients with suspected stable angina pectoris without coronary artery interventions, who showed a minimal to intermediate coronary artery diseases (a stenosis of 10 to 70% diameter as per QCA) in at least one natural coronary artery in coronary artery angiography or coronary artery CT.
3. Patients who gave their informed consent themselves in writing.
4. Patients who were treated with statin or lipid-lowering agents may participate in the study by changing the existing medicines.

Exclusion Criteria:

1. Patients with an intermediate (>30%) lesion on the left main coronary artery.
2. Patients diagnosed with acute coronary artery diseases (STEMI, NSTEMI, Unstable angina)
3. Patients who received percutaneous coronary intervention
4. Patients who have been diagnosed with stroke, transitory ischemic attack, and peripheral artery diseases.
5. Patients diagnosed with variant myocardial infarction
6. Patients with severe liver diseases or lung diseases and/or malignant tumor with life expectancy of less than 3 years
7. Patients with severe valvular heart disease
8. Patients who are hypersensitive or prohibited from using the active substance (Ezetimibe or Rosuvastatin) of the study medicines
9. Patients with cardiogenic shock
10. Pregnant women or women who are planning to get pregnant
11. Patients who are receiving hemodialysis or peritoneal dialysis or received renal transplantation due to end-stage renal failure
12. Patients who participated in other clinical studies within the past three months (except for non-interventional observation studies)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6356 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
The occurrence rates of the compound variables | Visit 5 (36month)
  The occurrence rates of the compound variables of all cause deaths, cardiac deaths, non-fatal myocardial infarction, non-fatal stroke, hospitalization due to unstable angina, and revascularization after taking the study medicine at the time of Visit 5 (36 month) were compared between groups

CONTACTS AND LOCATIONS:
Overall Officials: Sung-ho Her, MD.PhD, Principal Investigator — St Vincent's Hospital
Locations (1):
- St. Vincent's Hospital, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No